CLINICAL TRIAL: NCT05488340
Title: A Phase 2, Double-blind, Randomized, Active-controlled Evaluation of the Safety, Tolerability, Pharmacokinetics and Efficacy of LBP-EC01 in the Treatment of Acute Uncomplicated Urinary Tract Infection Caused by Drug Resistant E. Coli
Brief Title: A Study of LBP-EC01 in the Treatment of Acute Uncomplicated UTI Caused by Drug Resistant E. Coli (ELIMINATE Trial)
Acronym: ELIMINATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Locus Biosciences (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LBx-2001
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Urinary Tract Infections
Keywords: LBP-EC01; Urinary tract infection; E. coli; Bacteriophage; Phage; crPhage; Recombinant bacteriophage
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 - open label, Part 2 - blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1- Arm 4 (previously 1) (Experimental): Intraurethral (IU) LBP-EC01 on D1 and D2 with intravenous (IV) LBP-EC01 (1x10^11 PFU) and oral TMP/SMX on D1 through D3.
  Interventions: Drug: LBP-EC01 0.1 x IV dose; Drug: TMP/SMX
- Part 1- Arm 5 (previously 2) (Experimental): Intraurethral (IU) LBP-EC01 on D1 and D2 with intravenous (IV) LBP-EC01 (1x10^10 PFU) and oral TMP/SMX on D1 through D3.
  Interventions: Drug: LBP-EC01 0.01x IV Dose; Drug: TMP/SMX
- Part 1- Arm 6 (previously 3) (Experimental): Intraurethral (IU) LBP-EC01 on D1 and D2 with intravenous (IV) LBP-EC01 infusion (1x10^12 PFU) and oral TMP/SMX on D1 through D3.
  Interventions: Drug: LBP-EC01 IV Infusion Dose; Drug: TMP/SMX
- Part 2: LBP-EC01 (Experimental): LBP-EC01 given by dose regimen selected from Part 1. IU LBP-EC01 on D1 and D2 with IV LBP-EC01 (1x10^11 PFU) and oral TMP/SMX on D1 through D3.
  Interventions: Drug: LBP-EC01; Drug: TMP/SMX
- Part 2: Placebo (Placebo Comparator): Placebo given by dose regimen selected from Part 1. IU placebo on D1 and D2 with IV placebo and oral TMP/SMX on D1 through D3.
  Interventions: Drug: Placebo; Drug: TMP/SMX

INTERVENTIONS:
Drug: LBP-EC01 0.1 x IV dose — Intraurethral (IU) dose of two (2) x 6mL vials of LBP-EC01 (approximately 2x10^12 PFU) diluted in 188 mL of Lactated Ringer's solution on Day 1 and Day 2. Intravenous (IV) dose of 0.6mL of LBP-EC01 (approximately 1x10^11 PFU) diluted in 0.4mL of Lactated Ringer's solution given on Days 1 through Day 3.
  Other Names: 1x10^11 PFU IV dose
  Arms: Part 1- Arm 4 (previously 1)
Drug: LBP-EC01 0.01x IV Dose — Intraurethral (IU) dose of two (2) x 6mL vials of LBP-EC01 (approximately 2x10^12 PFU) diluted in 188 mL of Lactated Ringer's solution on Day 1 and Day 2. Intravenous (IV) dose of 0.06 mL of LBP-EC01 (approximately 1x10^10 PFU) diluted in 0.94 mL of Lactated Ringer's solution given on Days 1 through Day 3.
  Other Names: 1x10^10 PFU IV Dose
  Arms: Part 1- Arm 5 (previously 2)
Drug: LBP-EC01 IV Infusion Dose — Intraurethral (IU) dose of two (2) x 6mL vials of LBP-EC01 (approximately 2x10^12 PFU) diluted in 188 mL of Lactated Ringer's solution on Day 1 and Day 2. Intravenous infusion dose of 6mL of LBP-EC01 (approximately 1x10^12 PFU) diluted in 94 mL of Lactated Ringer's solution given over 2 hours on Days 1 through Day 3.
  Other Names: 1x10^12 PFU IV Infusion Dose
  Arms: Part 1- Arm 6 (previously 3)
Drug: Placebo — Dose regimen selected from Part 1 of placebo (Tris buffer).
  Arms: Part 2: Placebo
Drug: LBP-EC01 — Dose regimen selected from Part 1 of LBP-EC01 (1x10^10 - 1x10^13 PFU) per dose.
  Arms: Part 2: LBP-EC01
Drug: TMP/SMX — TMP/SMX (160 mg trimethoprim and 800 mg sulfamethoxazole) given orally BID on Days 1 through 3.

SUMMARY:
This is a Phase 2 superiority study of LBP-EC01, a recombinant bacteriophage cocktail, with an initial open-label 3-arm pharmacokinetic (PK) lead-in portion of 30 patients to evaluate the optimal dosing regimen to be used in the subsequent 288 patient blinded portion of the study which will be randomized 1:1 comparing LBP-EC01 + antibiotic versus placebo + antibiotic in patients with a history of prior urinary tract infection (UTI) cased by E. coli. All patients will be required to have an active acute uncomplicated UTI at baseline.

DETAILED DESCRIPTION:
This study will consist of two parts.

Part 1 - Dose regimen selection: An open-label, 30 patient, 3-arm PK assessment of: Arm 4 (previously 1): LBP-EC01 (approximately 2×10^12 PFU) given by IU administration on D1 and D2 and LBP-EC01 (approximately 1×10^11 PFU) IV given as a 1 milliliter (mL) bolus QD from D1 through D3 concomitantly with oral trimethoprim/sulfamethoxazole (TMP 160mg/SMX 800mg) BID from D1 through D3 (6 doses); Arm 5 (previously 2): LBP-EC01 (approximately 2×10^12 PFU) given by IU administration on D1 and D2 and LBP-EC01 (approximately 1×10^10 PFU) IV given as a 1 mL bolus QD from D1 through D3 concomitantly with oral TMP/SMX BID from D1 through D3 (6 doses); Arm 6 (previously 3): LBP-EC01 (2×10^12 PFU) given by IU administration on D1 and D2 and LBP-EC01 (approximately 1×10^12 PFU) IV given as a 100 mL IV infusion over 2 h on D1 through D3 concomitantly with oral TMP/SMX BID from D1 through D3 (6 doses).

Part 2 - Efficacy, Safety, Tolerability and Pharmacokinetics: A blinded, 288 patient, 1:1 randomized evaluation of the Arm 4 dose regimen, selected from Part 1, versus placebo + antibiotic (TMP/SMX -160 mg TMP and 800 mg SMX) given orally BID on Days 1 through 3.

ELIGIBILITY:
Inclusion Criteria:

* History of UTI in the past 12 months and prior or current uUTI caused by AMR E. coli (as single pathogen or part of polymicrobial infection where E. coli is the predominant pathogen). Please note that the current infection can be used to meet the requirement of AMR E. coli documentation.
* Able to supply a mid-stream, clean catch urine sample for microbiological analysis.
* Active acute uUTI infection defined by:

  a. Evidence of pyuria: i. >10 white blood cell (WBC)/mL3 on microscopic evaluation of spun, clean, mid-stream urine specimen or >3 WBC/high power field on unspun clean, mid-stream urine specimen, AND/OR ii. Dipstick analysis of a clean, mid-stream urine specimen positive for leukocytes, AND b. At least 2 of the following signs or symptoms of UTI: dysuria, urinary frequency, urinary urgency, or suprapubic pain
* Willing to comply with all aspects of study design including study restrictions, blood, urine, and stool sampling, and scheduled study visits.
* All sexually active female patients of childbearing potential must use highly effective contraception during the study and until 2 weeks after the last dose of study drug treatment.
* Agrees to STOP continuous low dose antimicrobial prophylaxis and/or will maintain the same practices for post-coital antimicrobial prophylaxis to prevent UTI, as during the prior 12-months, for the entire study duration (throughout the 6-month follow-up period or study discharge).
* Agrees to not use any prescription or non-prescription medication for the microbiological or symptomatic treatment of the presenting acute uUTI for the first 10 days of the study.
* Capable of providing their own signed informed consent form (ICF) prior to any study-related procedures being performed.
* If participating in Part 1 of the study, agrees to fast for ≥2 h prior to first dose of study drug on Day 1/Visit 1 except for drinking 240 mL of water with study drug administration.

Exclusion Criteria:

* Signs or symptoms of systemic illness such as fever greater than 38° Centigrade/ Celsius, shaking chills, or other clinical manifestations suggestive of complicated UTI.
* Treatment with other antibacterial drugs including those that are effective for treatment of the acute uUTI or prevention of recurrent UTI in the 5 days prior to Screening unless the recovered pathogen demonstrates resistance to the initial antibiotic and clinical symptoms persist. In postmenopausal women vaginal estrogen replacement therapy is permitted so long as patient meets all other eligibility criteria, that the dose and regimen has be stable for > 3 months from Screening (D1/V1), and that there is no planned change to therapy through the 6-month follow-up period or study discontinuation.
* Clinical symptoms for more than 5 days before Screening.
* Presence of indwelling urinary bladder catheters, urinary tract anatomical abnormalities that increase UTI risk or lead to a post void residual (PVR) urine volume > 150mL, poorly controlled diabetes mellitus (diagnosed but is not being treated/managed by a physician's care or HbA1c >8), current symptomatic or larger than 5mm renal calculi, or advanced renal dysfunction (determined by eGFR < 45 mL/min/1.73 m2). Patients with vaginal prolapse beyond the hymen with Valsalva (e.g., when coughing).
* Individuals considered to be immunocompromised.
* Clinically significant serious unstable physical illness that in the investigator's opinion prevents patient from completing the study or prevents interpretation or resolution of clinical symptoms.
* Pregnant or nursing women.
* Exposure to any investigational drugs or other phage therapy 30 days prior to Screening (D1/V1) or prior to participation in this study. Patients who participate in Part 1 are not eligible for participation in Part 2.
* Allergies to excipients of the study drug or antibiotics.
* History of autonomic dysreflexia.
* History of intravenous (IV) drug abuse or is currently using or has positive results for drugs of abuse at screening.
* Patients who reside in a long-term care facility.
* Suspected or confirmed acute coronavirus disease 2019 (COVID-19) or recent COVID-19 infection with ongoing symptoms.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 318 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Part 1: Levels of LBP-EC01 in urine and blood measured by quantitative plaquing assay across the treatment period and over 48 h after the last dose | Day 1 to Day 5
  The regimen for LBP-EC01 when used concomitantly with TMP/SMX which optimizes pharmacokinetics (PK) for LBP-EC01 will be selected.
Part 2: Proportion of patients with resolution of clinical symptoms and microbiologic response of uUTI caused by drug resistant E. coli as defined at Day 10 test of cure (TOC). | Day 10
  The efficacy of LBP-EC01 when used concomitantly with TMP/SMX compared to placebo when used concomitantly with TMP/SMX on resolution of acute uUTI clinical symptoms and demonstration of microbiologic response (CCMR) of acute uUTI caused by drug resistant E. coli will be assessed.

SECONDARY OUTCOMES:
Part 1: Number of patients with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 to Day 34
  The safety and tolerability of LBP-EC01 when given with TMP/SMX will be assessed.
Part 1: Number of patients with immunogenicity | Baseline Day 1 to Day 2, Day 5, Day 10, Day 34/Early Termination [ET]) post-hoc
  The immunogenicity of LBP-EC01 by measuring neutralizing antibody (NAb) levels will be assessed.
Part 2: Proportion of patients with antimicrobial drug resistant (AMR) E. coli achieving maintenance of combined clinical and microbiologic response (CCMR) at Day 21. | Day 21
  The impact of LBP-EC01 when used concomitantly with TMP/SMX compared to placebo when used concomitantly with TMP/SMX on maintenance of CCMR success in those randomized patients with AMR E. coli uUTI demonstrating an initial response will be assessed.
Part 2: Proportion of patients with CCMR of uUTI caused by E. coli at Day 10/TOC. | Day 10
  The efficacy of LBP-EC01 when used concomitantly with TMP/SMX compared to placebo when used concomitantly with TMP/SMX, on CCMR of uUTI caused by E. coli (irrespective of drug resistant status) will be assessed.
Part 2: Proportion of patients with CCMR of uUTI caused by multi-drug resistant (MDR) E. coli at Day 10/TOC. | Day 21
  The impact of LBP-EC01 when used concomitantly with TMP/SMX compared to placebo when used concomitantly with TMP/SMX on CCMR in patients with uUTI caused by MDR E. coli at Day 10/TOC.
Part 2: Proportion of patients with MDR E. coli achieving maintenance of CCMR at Day 21. | Within the 6-month follow-up period
  The impact of LBP-EC01 when used concomitantly with TMP/SMX compared to placebo when used concomitantly with TMP/SMX on the maintenance of CCMR in patients with uUTI caused by MDR E. coli at Day 21.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kim, Study Director — Locus Biosciences
Locations (12):
- United States (12):
  - Research Site 138, Fresno, California
  - Research Site 131, Lancaster, California
  - Research Site 123, Los Angeles, California
  - Research Site 125, Montebello, California
  - Research Site 137, San Diego, California
  - Research Site 126, Tustin, California
  - Research Site 102, Doral, Florida
  - Research Site 140, Jensen Beach, Florida
  - Research Site 103, Miami, Florida
  - Research Site 149, Miami, Florida
  - Research Site 120, Boston, Massachusetts
  - Research Site 118, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim P, Sanchez AM, Penke TJR, Tuson HH, Kime JC, McKee RW, Slone WL, Conley NR, McMillan LJ, Prybol CJ, Garofolo PM. Safety, pharmacokinetics, and pharmacodynamics of LBP-EC01, a CRISPR-Cas3-enhanced bacteriophage cocktail, in uncomplicated urinary tract infections due to Escherichia coli (ELIMINATE): the randomised, open-label, first part of a two-part phase 2 trial. Lancet Infect Dis. 2024 Dec;24(12):1319-1332. doi: 10.1016/S1473-3099(24)00424-9. Epub 2024 Aug 9. PMID 39134085